CLINICAL TRIAL: NCT05006859
Title: Wheelchair Positioning and Neuromuscular Diseases Database (Retrospective and Prospective)
Brief Title: Wheelchair Positioning and Neuromuscular Diseases
Acronym: BDD-POSIT-MNM
Status: Recruiting | Type: Observational
Sponsor: Groupement Hospitalier Intercommunal du Vexin (Other)
Collaborators: Association Française contre les Myopathies (AFM), Paris (Other)
Responsible Party: Sponsor
Other Study IDs: GHIV0321
Record Dates: First submitted 2021-08-11; First posted 2021-08-16 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Neuromuscular Diseases
Keywords: Neuromuscular disease; Postural wheelchair disorders; Wheelchair positioning; Pain
MeSH Terms: conditions — Neuromuscular Diseases; Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Cohorte — Assessment of postural wheelchair disorders, as well as PW pain, and pressure ulcers associated with sitting
  Other Names: Questionnaire

SUMMARY:
This database will describe sitting postural control in wheelchair, as well as PW pain, and pressure ulcers associated with sitting, in patients with neuromuscular disease (NMD).

DETAILED DESCRIPTION:
Neuromuscular diseases are genetic diseases of the muscle or its innervation (nerve connection) causing respiratory, cardiac and especially motor difficulties which may require use of wheelchair. However there is no standardized positioning protocol, so it seems interesting to us to study wheelchair positioning in neuromuscular diseases).

The purpose of this study is to describe sitting posture in the wheelchair in patients with neuromuscular disease, pain associated with using the wheelchair, but also to assess the effectiveness of the recommended equipment making the same evaluations in follow-up consultation (a few months after receipt of the prescribed TAP).

Posture is assessed by the tool: Measurement of Postural Control in Seated Postural Control Measure for Adults 2.0 (SPCMA 2.0), which is a validated tool.

Pain is assessed by a Simple Verbal Scale or by a Visual Analog Scale. This database could allow providing guidelines of good practice, for wheelchair positioning for patients with neuromuscular disease.

ELIGIBILITY:
Inclusion Criteria :

* Patient with neuromuscular disease
* Written informed consent (IC) obtained
* Adult patients (> 18 years) Or
* Adults under guardianship who has given theirs oral consent and guardian's consent obtained Or
* Childs who has given theirs oral consent and parents' consent obtained
* Wheelchair user

Exclusion Criteria :

• Patient not seen in positioning consultation by N. Pellegrini and / or E. Dupitierr

Min Age: 8 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with neuromuscular disease, using Wheelchair, seen in positioning consultation by N. Pellegrini and / or E. Dupitier
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-05-17 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Description of postural wheelchair disorders in the neuromuscular disease population | At the beginning and the end of the study, an average of 6 months
  Measurement of Posture by the tool: Measurement of Postural Control in Seated Postural Control Measure for Adults 2.0 (SPCMA 2.0) score (0 = normal, 1 = mild, 2 = moderated and 3 = severe)

SECONDARY OUTCOMES:
Comparison of pain associated with using the wheelchair | At the beginning and the end of the study (before positioning equipment and few months after use), an average of 6 months
  Assessment of initial pain (before positioning equipment) and pain after positioning equipment.
  Pain is assessed by a Simple Verbal Scale or by a Visual Analog Scale (0 to 10) (0 = no pain and 10 is the strongest pain)
Assessment of the incidence of pressure ulcers associated with sitting in NMD | At the beginning and the end of the study (before positioning equipment and few months after use), an average of 6 months
  Observation of the topography and the stage of ulcers associated with sitting
Assessment of the proportion of technical postural aids prescribed for patients who accept the positioning equipment | At the end of the study, an average of 6 months
  Counts of the numbers of technical postural aids prescribed during consultation
Assessment of the technical postural aids efficacy | At the beginning and the end of the study (before positioning equipment and few months after use), an average of 6 months
  Comparison of Postural Control in Seated Postural Control Measure for Adults 2.0 (SPCMA 2.0) score before and after using of technical postural aids (0 = normal, 1 = mild, 2 = moderated and 3 = severe)

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Pellegrini, Principal Investigator — Groupement Hospitalier Intercommunal du Vexin
Locations (2):
- France (2):
  - Groupement Hospitalier Intercommunal du Vexin / Site d'Aincourt - Pôle Soins de Suite et de Réadaptation spécialisés, Aincourt
  - Clinique du Positionnement de l'AFM, Évry